CLINICAL TRIAL: NCT00947817
Title: Impact of Endothelial Cell Activation and Modifications of Haemostasis Induced by Infective Endocarditis on the Risk of Embolism.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008 07; 2008-A00114-51
Record Dates: First submitted 2009-01-15; First posted 2009-07-28 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2010-05

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient (Experimental)
  Interventions: Other: ULTRASONOGRAPHY trans-esophageal and trans-thoracic , blood test and clinic test
- control (Other)
  Interventions: Other: ULTRASONOGRAPHY trans-esophageal and trans-thoracic , blood test and clinic test

INTERVENTIONS:
Other: ULTRASONOGRAPHY trans-esophageal and trans-thoracic , blood test and clinic test

SUMMARY:
Prospective study including all the consecutive patients admitted at the Department of Cardiology, Timone Hospital wih a definite diagnosis of IE according to the modified Duke criteria. The period of inclusion will be for 24 months. Eighty patients and age-matched control subject will be included. Primary end point are EE occurring during the antimicrobial treatment and secondary end points will be 6-month mortality, vegetation length and the impact of antimicrobial treatment on inflammation-induced procoagulant changes and endothelial cell activation.

ELIGIBILITY:
Inclusion Criteria:

* All the patients presenting certain diagnosis of infectious endocardite according to the criteria of modified Duke

Exclusion Criteria:

* Age < 18 years
* Pregnancy and feeding
* Health not allowing to give the assent
* Innate abnormalities of the haemostasis
* More than a week before the inclu antibiothérapie adapted begun

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2008-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Embolic events occurring during the antimicrobial treatment a | 30 months

SECONDARY OUTCOMES:
Will be 6-month mortality, vegetation length and the impact of antimicrobial treatment on inflammation-induced procoagulant changes and endothelial cell activation. | 30months

CONTACTS AND LOCATIONS:
Overall Officials: franck thuny, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Département de Cardiologie, Unité Valvulopathies et Insuffisance Cardiaque, Hôpital de la Timone,, Marseille, Paca, France